CLINICAL TRIAL: NCT06335225
Title: Establishment of Precise Nutrition Management Scheme for Patients With Prediabetes Based on Nutrigenomics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Ma Xiao, Director of health examination center department, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-NHLHCRF-YXHZ-ZRMS-06
Record Dates: First submitted 2024-03-15; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Prediabetes
Keywords: Prediabetes; Nutrigenomics; Nutritional intervention
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precise nutrition group (Experimental)
  Interventions: Behavioral: Precise nutritional intervention
- Control group (Active Comparator)
  Interventions: Behavioral: Conventional nutritional intervention

INTERVENTIONS:
Behavioral: Precise nutritional intervention — Diabetic precision nutrition prescription based on the results of nutrigenomics.
  Arms: Precise nutrition group
Behavioral: Conventional nutritional intervention — Conventional diabetes nutrition prescription.
  Arms: Control group

SUMMARY:
With the aging of population and the change of lifestyle, the prevalence of prediabetes is increasing year by year. Nutritional factors are one of the important environmental factors in the occurrence and development of abnormal glucose metabolism. The medical nutritional treatment of diabetes is recommended as the cornerstone of diabetes treatment by various guidelines. With the development of nutrigenomics, it has been found that genes related to the absorption, metabolism, distribution and excretion of various nutrients are related to diabetes. This study intends to conduct precision nutrition intervention for prediabetic patients based on nutritional genes, and evaluate the effectiveness and safety of these nutritional interventions.

ELIGIBILITY:
Inclusion Criteria:

1. OGTT: 6.1 mmol/L ≤ fasting plasma glucose < 7.0 mmol/L and（or）7.8 mmol/L ≤ 2 hour plasma glucose < 11.1 mmol/L and (or) 5.7% ≤ HbA1c< 6.5%.
2. 18 ≤ Age <70.

Exclusion Criteria:

1. Patients who can be diagnosed with diabetes mellitus.
2. Patients applying antidiabetic drugs, glucocorticoids, and other drugs that have an effect on blood glucose.
3. Females during pregnancy or lactation.
4. Patients with gastrointestinal disorders, psychiatric disorders, autoimmune disorders, tumors, etc.
5. Patients with acute cardiovascular and (or) cerebrovascular diseases within 6 months prior to study participation.
6. Patients with hepatic dysfunction (ALT, AST, or total bilirubin ≥ 2 times the upper limit of normal), renal dysfunction (creatinine > the upper limit of normal), and cardiac dysfunction (NYHA class III and IV).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | week 0, week 12, week 24

SECONDARY OUTCOMES:
Concentration of fasting plasma glucose | week 0, week 12, week 24
Concentration of 2-hour plasma glucose | week 0, week 24
Concentration of fasting insulin | week 0, week 12, week 24
Concentration of fasting C peptide | week 0, week 12, week 24
Concentration of TC, TG, LDL-C, and HDL-C | week 0, week 12, week 24
Concentration of ALT, AST, TBIL | week 0, week 12, week 24
Concentration of creatinine | week 0, week 12, week 24
BMI | week 0, week 4, week 8, week 12, week 16, week 20, week 24
  BMI (kg/m^2) =body weight/(height)^2
Waist hip ratio | week 0, week 4, week 8, week 12, week 16, week 20, week 24
  Waist hip ratio = waist circumference/hip circumference

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China